CLINICAL TRIAL: NCT05556408
Title: High-Resolution Solid-State Manometry of the Effect of Succinylcholine on Barrier Pressure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Yanting Cao, PhD, China-Japan Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: the Effect of Succinylcholine
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: the Effect of Succinylcholine on Barrier Pressure
Keywords: lower esophageal sphincter; intragastric pressure; succinylcholine
MeSH Terms: interventions — Succinylcholine; Propofol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-Resolution Solid-State Manometry (Other): Before catheterization, the patients were monitored by pulse oximetry, electrocardiogram, automatic noninvasive arterial blood pressure and bispectral index (BIS). Before the insertion of the manometric catheter an intravenous cannula was inserted. The manometric catheter was placed through the nose until the pressure from the lower esophageal sphincter to the stomach could be recorded. After confirming the position of the catheter, the catheter was taped to the nose.
  Interventions: Drug: Succinylcholine

INTERVENTIONS:
Drug: Succinylcholine — 1.5mg/kg was given intravenously
  Other Names: propofol

SUMMARY:
The lower esophageal sphincter（LES）plays a key role in preventing regurgitation and aspiration. The pressure of LES partly comes from striated muscles derived from the crural portion of the diaphragm. The effect of succinylcholine on esophagogastric junction during anesthesia induction is not clear. We conducted a prospective interventional study on the effect of succinylcholine on the barrier pressure (BrP) of the esophagogastric junction.

DETAILED DESCRIPTION:
14 patients participated in the study. Propofol and succinylcholine were used for anesthesia induction. High-resolution solid-state manometry (HRM) was used to monitor the changes of the LES pressure and the intragastric pressure (IGP).The administration of propofol could significantly increase the LES pressure during end expiration and during inspiration. The application of succinylcholine had no effect on the LES pressure during end expiration, but significantly reduced the LES pressure during inspiration. Propofol had no effect on BrP. After the application of succinylcholine, BrP decreased significantly during inspiration.

Propofol significantly increased the LES pressure. Succinylcholine significantly reduced the pressure of LES and BrP during inspiration.

ELIGIBILITY:
Exclusion criteria：patients who classified as American Society of Anesthesiologists classification system (ASA) II were included. Patients were included in the study if they had on history of diabetes, pharynx and digestive diseases.

Exclusion criteria：currently pregnant or breastfeeding, a body mass index (BMI) over 30 kg/m2. All patients underwent preoperative preparation according to clinical routine and did not give preoperative drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
pressure of lower esophageal sphincter | 15 minutes
  On the isocontour plots, the esophageal sphincter can be located as abrupt transitions in the pressure pattern (Fig. 2). The proximal edge of the LES was defined by sudden transition to the intra-esophageal pressure, and the distal edge was defined by sudden transition to the IGP. The pressure of the LES measured during end expiration was defined as the pressure of intrinsic sphincter to avoid the influence from the rural component of the LES. The rural component of the LES was defined as the highest pressure point at the esophagogastric junction during inspiration.
pressure of intragastric | 15 minutes
  IGP was measured at 2 cm below the crural diaphragmatic component of the LES

IPD SHARING:
Plan to Share IPD: No